CLINICAL TRIAL: NCT02891291
Title: Optical Tomographic Scanner for Skin Lesions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 201604078RINB
Record Dates: First submitted 2016-09-01; First posted 2016-09-07 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Skin Cancer, Benign Skin Tumor, Inflammatory Skin Disease
Keywords: optical coherence tomography
MeSH Terms: conditions — Skin Neoplasms; Dermatitis

STUDY DESIGN:
Biospecimen Retention: Samples Without DNA — skin tissue sample
Oversight: Data Monitoring Committee: No

SUMMARY:
Optical coherence tomography is technology widely used in medicine. In this study, the investigators will use an optical tomographic scanner to scan skin tissue image.

DETAILED DESCRIPTION:
The investigators will use optical tomographic scanner to scan skin specimen and obtain tissue images. Part of skin specimen obtained from skin biopsy or surgery will be scanned.

ELIGIBILITY:
Patient who receive skin biopsy or surgery due to skin cancers, benign skin diseases, or inflammatory skin diseases.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient's age are between 20 to 100 years old. Patients who receive skin biopsy or surgery at Department of Dermatology, National Taiwan University Hospital, Taiwan.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Skin tissue image obtained. | 1 week
  Part of the skin specimen from surgery or biopsy will be scanned.

SECONDARY OUTCOMES:
Skin histopathology | 2 week
  The skin specimen will be stained with hematoxylin and eosin. Histopathological pictures (or findings) will be obtained and correlate with the scanned images.

CONTACTS AND LOCATIONS:
Overall Officials: JENGWEI TJIU, MDPHD, Principal Investigator — NTUH
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No
No plan to share data.